CLINICAL TRIAL: NCT04522713
Title: Single-Arm Feasibility Study of a Transdiagnostic Course for Common Mental Health Problems in Primary Care
Brief Title: A Transdiagnostic Course for Common Mental Health Problems in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erland Axelsson, Principal Investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-04816
Record Dates: First submitted 2020-08-10; First posted 2020-08-21 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Depression; Anxiety
Keywords: Transdiagnostic; Primary care; Feasibility
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective single-group cohort study
Masking Description: Psychological intervention, self-report outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Large-group transdiagnostic course (Experimental): 6 weekly structured transdiagnostic large-group course sessions which focus on evidence-based strategies to reduce psychiatric symptoms and increase wellbeing
  Interventions: Behavioral: Behavioral activation, evidence-based sleep strategies including sleep restriction, exposure-based strategies, promotion of physical activity and recuperating activities, psychoeducational material

INTERVENTIONS:
Behavioral: Behavioral activation, evidence-based sleep strategies including sleep restriction, exposure-based strategies, promotion of physical activity and recuperating activities, psychoeducational material — Primarily standard cognitive-behavioral strategies to reduce common psychiatric symptoms

SUMMARY:
This study investigates the feasibility of a transdiagnostic course that is intended to work for a large variety of patient groups with clinically significant depression or anxiety in primary care. This is a prospective single-group study where 68 adults with clinically significant symptoms of depression or general anxiety, and up to 25 adults with subclinical symptoms, attend up to 6 weekly structured large-group course sessions which focus on evidence-based strategies to reduce psychiatric symptoms and increase wellbeing. If necessary, due to the covid-19 pandemic, the course will be held online.

DETAILED DESCRIPTION:
Background:

Depression and the common anxiety disorders are highly prevalent and associated with disability and reduced quality of life. There is reason to believe that the majority of these patients are found in primary care. Official Swedish guidelines dictate that primary care clinics are responsible for treating mild to moderate cases, but access to treatment is limited. Transdiagnostic psychological interventions have been found to be efficacious for anxiety and mood disorders, and require a relatively rudimentary pre-treatment assessment. A large-group transdiagnostic course based on cognitive-behavioral principles may constitute an effective use of limited resources to improve access to treatment, and offer a sufficiently effective intervention, for most primary care patients with mild to moderate mental health problems.

Aim:

To investigate the feasibility and preliminary efficacy of a large-group transdiagnostic intervention for depression and clinically significant anxiety in Swedish primary care.

Design:

This is a prospective single-group feasibility study where 68 adults with clinically significant symptoms of depression or anxiety, and up to 25 adults with subclinical symptoms, are recruited from Liljeholmen primary care clinic, Stockholm, and offered 6 weekly structured transdiagnostic large-group course sessions which focus on evidence-based strategies to reduce psychiatric symptoms and increase wellbeing. If necessary, due to the covid-19 pandemic, the course will be held online. The primary outcome is patient satisfaction. Secondary outcomes include within-group effects on psychiatric symptoms (response rates), adherence rates, need for additional treatment, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* At least 8 points on the GAD-7 or 10 points on the PHQ-9 (N=68; up to 25 subclinical participants may also take part in the study)
* At least 18 years old

Exclusion Criteria:

* At least one severe mental health problem such as suicidal ideation, a bipolar disorder, or psychosis
* Non-stable antidepressant medication (dosage changed during the past 6 weeks)
* Planned absence for 2 weeks or more of the intended treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erland Axelsson, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Liljeholmen primary care clinic, Stockholm
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: No
We are willing to consider reasonable requests for individual participant data (IPD) and to consult the responsible parties accordingly. However, we do not expect to be granted permission to share IPD as long as, under Swedish and European Union (EU) data protection and privacy legislation, the IPD constitutes personal data meaning that it is possible to, using the study database, link the IPD to an identifiable living natural person.

REFERENCES:
- [Derived] Kolaas K, Berman AH, Hedman-Lagerlof E, Zakrevska A, Epstein M, Hammarberg SAW, Axelsson E. Feasibility of a video-delivered mental health course for primary care patients: a single-group prospective cohort study. BMC Prim Care. 2023 Jan 23;24(1):28. doi: 10.1186/s12875-023-01989-8. PMID 36690940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We intended to recruit 68 participants with clinically significant depression or anxiety, and up to 25 participants with subclinical depression and anxiety. When the target of 68 clinical participants had been met, the remaining scheduled eligibility interviews were completed for ethical reasons, which resulted in a final clinical sample size of 70. By that time, 21 subclinical participants had been enrolled, which resulted a total sample size of 91.
Pre-assignment Details: All participants were enrolled in the course.
Groups:
- Large-group Transdiagnostic Course: All participants took part in the same intervention, and were analyzed as one group. There were no subgroups receiving separate interventions.
  6 weekly structured transdiagnostic large-group course sessions which focus on evidence-based strategies to reduce psychiatric symptoms and increase wellbeing
  Behavioral activation, evidence-based sleep strategies including sleep restriction, exposure-based strategies, promotion of physical activity and recuperating activities, psychoeducational material: Primarily standard cognitive-behavioral strategies to reduce common psychiatric symptoms
Period: Overall Study
Arm/Group | Large-group Transdiagnostic Course
Started | 91
Completed (Completed the post-course assessment after week 6) | 86
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: In this feasibility study, in accordance with the preregistered plan, no distinction between clinical and subclinical participants was done except for the auxilliary preliminary efficacy analyses. All 91 participants were recruited via the same pathway, followed the same protocol, and were considered part of the same cohort.
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 91
University education [Count of Participants; unit: Participants] | 71
Employment [Count of Participants; unit: Participants]
  Working full-time | 55
  Working part-time (< 90%) | 11
  Unemployed | 3
  Retired | 3
  Student | 9
  Other | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Satisfaction With Treatment
Description: Preregistered target: mean Client Satisfaction Questionnaire (CSQ-8) score of at least 22. Theoretical range: 8-32, higher score indicates higher satisfaction. This sum score is based on 8 items, each scored 1-4. The original preregistered range of 7-28 was an erratum.
Time Frame: Post-course assessment (immediately after the course, completed within 45 days)
Population: The trial included 91 participants: 70 clinical, and 21 subclinical. Of these, 86 (66 + 20) completed the CSQ-8 at the post-course assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 86
score on a scale
  Pooled sample (primary) | 22 (4)
  Clinical subsample: number analyzed (Participants) | 66
  Clinical subsample | 21 (4)
  Subclinical subsample: number analyzed (Participants) | 20
  Subclinical subsample | 23 (3)
  Participants without previous experience of psychological treatment: number analyzed (Participants) | 34
  Participants without previous experience of psychological treatment | 23 (4)
  Participants with previous experience of psychological treatment: number analyzed (Participants) | 52
  Participants with previous experience of psychological treatment | 21 (4)

2. Secondary Outcome: Adherence Operationalized as the Average Number of Attended Lectures
Description: Attendance, i.e., participation in the course, registered once each week, after each course date, by a clinician during the course period
Time Frame: From week 1 to week 6
Measure: Mean (Standard Deviation); unit: lectures attended
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 91
lectures attended | 5.0 (1.6)

3. Secondary Outcome: Number of Participants With Clinically Significant Improvement in Symptoms of Depression
Description: Preregistered target: At least 1/3 patients reporting a clinically significant improvement in symptoms of depression. Dichotomous outcome based on the Patient Health Questionnaire 9 (PHQ-9, theoretical range: 0-27, higher score indicates more symptoms of depression). Clinically significant improvement implied a reduction of at least 6 points on the PHQ-9 in combination with a post-course score below 10.
Time Frame: Pre-course assessment (within 2 weeks before the course) to post-course assessment (immediately after the course, completed within 45 days)
Population: For depression symptoms, only those who had a score of at least 10 on the PHQ-9 at baseline could potentially be classified as clinically significant improved. This was done to ensure that the clinical cut-off was not too liberal and also that all participants scored in the clinical range at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 46
Participants | 22

4. Secondary Outcome: Number of Participants With Clinically Significant Improvement in General Anxiety
Description: Preregistered target: At least 1/3 patients reporting a clinically significant improvement in general anxiety. Dichotomous outcome based on the GAD-7 (theoretical range: 0-21, higher score indicates more general anxiety). Clinically significant improvement implied a reduction of at least 5 points on the GAD-7 in combination with a post-course score below 8.
Time Frame: as for outcome 3
Population: For general anxiety, only those who had a score of at least 8 on the GAD-7 at baseline could potentially be classified as clinically significant improved. This was done to ensure that the clinical cut-off was not too liberal and also that all participants scored in the clinical range at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 46
Participants | 27

5. Secondary Outcome: Number of Participants With Problematic Lifestyle Behaviors
Description: Lifestyle behaviors were measured using the Lifestyle Behaviors Questionnaire (LBQ) which comprises 11 items that cover tobacco use, alcohol use, physical activity and diet. Dichotomous risky lifestyle behavior variables were derived from the LBQ in terms of: "At least one unhealthy lifestyle behavior", "Daily smoking", "Binge drinking more than once a month OR more than 9/14 (w/m) glasses/week", "Insufficient physical activity, less than 150 minutes/week", and "Notably unhealthy dietary habits (diet index 0-4)". Risky lifestyle behavior was defined as daily smoking, binge drinking of 4/5 (women/men) drinks at one occasion more than once a month and/or more than 9/14 (women/men) standard glasses of alcohol weekly, insufficient physical activity (<150 minutes/week) or significantly unhealthy diet habits (a score of 0-4 on a diet index in the questionnaire, ranging from 0-12).
Time Frame: as for outcome 3
Population: 86/91 participants completed the post-course assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 91
Participants
  Pre-course: At least one unhealthy lifestyle behavior | 40
  Post-course: At least one unhealthy lifestyle behavior: number analyzed (Participants) | 86
  Post-course: At least one unhealthy lifestyle behavior | 36
  Pre-course: Daily smoking | 2
  Post-course: Daily smoking: number analyzed (Participants) | 86
  Post-course: Daily smoking | 2
  Pre-course: Binge drinking more than once a month OR more than 9/14 (w/m) glasses/week | 17
  Post-course: Binge drinking more than once a month OR more than 9/14 (w/m) glasses/week: number analyzed (Participants) | 86
  Post-course: Binge drinking more than once a month OR more than 9/14 (w/m) glasses/week | 15
  Pre-course: Insufficient physical activity, less than 150 minutes/week | 22
  Post-course: Insufficient physical activity, less than 150 minutes/week: number analyzed (Participants) | 86
  Post-course: Insufficient physical activity, less than 150 minutes/week | 22
  Pre-course: Notably unhealthy dietary habits (diet index 0-4) | 11
  Post-course: Notably unhealthy dietary habits (diet index 0-4): number analyzed (Participants) | 86
  Post-course: Notably unhealthy dietary habits (diet index 0-4) | 15

6. Secondary Outcome: Number of Adverse Events
Description: Weekly question: "Since the last assessment, have you experienced any adverse event, side effect, or unwanted effect of your participation in this study?"
Time Frame: From week 1 to week 6
Population: 86/91 participants completed the post-course assessment at week 6
Measure: Number; unit: adverse events reported
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 86
adverse events reported | 9

7. Secondary Outcome: Percentage of Patients in Need of Additional Clinical Intervention
Description: Clinical interview
Time Frame: Post-course assessment (within 45 days after the course)
Population: 81/91 completed the post-course interview
Measure: Count of Participants; unit: Participants
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 81
Participants | 44

8. Secondary Outcome: Change in Mean Symptoms of Depression From Pre- to Post-Course Assessment
Description: Patient Health Questionnaire 9 (PHQ-9, theoretical range: 0-27, higher score indicates more symptoms of depression). Efficacy outcomes based on linear mixed models.
Time Frame: as for outcome 3
Population: 70 clinical, 21 subclinical
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 91
units on a scale
  Clinical subsample: number analyzed (Participants) | 70
  Clinical subsample | -4.8 [-6.1 to -3.4]
  Subclinical subsample: number analyzed (Participants) | 21
  Subclinical subsample | -1.5 [-2.8 to -1.5]

9. Secondary Outcome: Change in Mean General Anxiety From Pre- to Post-Course Assessment
Description: GAD-7 (theoretical range: 0-21, higher score indicates more general anxiety). Efficacy outcomes based on linear mixed models.
Time Frame: as for outcome 3
Population: 70 clinical, 21 subclinical
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 91
units on a scale
  Clinical subsample: number analyzed (Participants) | 70
  Clinical subsample | -3.8 [-5.0 to -2.6]
  Subclinical subsample: number analyzed (Participants) | 21
  Subclinical subsample | -1.2 [-2.3 to -0.6]

10. Secondary Outcome: Change in Mean Perceived Stress From Pre- to Post-Course Assessment
Description: Perceived Stress Scale, 10-item version (PSS-10, theoretical range: 0-40, higher score indicates more perceived stress). Efficacy outcomes based on linear mixed models.
Time Frame: as for outcome 3
Population: 70 clinical, 21 subclinical
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 91
units on a scale
  Clinical subsample: number analyzed (Participants) | 70
  Clinical subsample | -3.3 [-4.6 to -1.9]
  Subclinical subsample: number analyzed (Participants) | 21
  Subclinical subsample | -1.5 [-4.2 to 1.2]

11. Secondary Outcome: Change in Mean Disability From Pre- to Post-Course Assessment
Description: World Health Organization Disability Assessment Schedule 2.0 (WHODAS-2, theoretical range: 0-100, higher score indicates more disability). Efficacy outcomes based on linear mixed models.
Time Frame: as for outcome 3
Population: 70 clinical, 21 subclinical
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Large-group Transdiagnostic Course
Number analyzed (Participants) | 91
units on a scale
  Clinical subsample: number analyzed (Participants) | 70
  Clinical subsample | -4.1 [-7.1 to -1.1]
  Subclinical subsample: number analyzed (Participants) | 21
  Subclinical subsample | 0.4 [-4.3 to 5.1]

ADVERSE EVENTS:
Time Frame: 6-week course period
Description: At the post-course assessment, we assessed adverse events using free-text items where the respondent could report up to three adverse events, describe these in free text, and rate how much each adverse event had affected them negatively at the time it occurred, and still affected them negatively at the post-course assessment.
Arm/Group | Large-group Transdiagnostic Course
All-Cause Mortality (participants affected / at risk) | 0/91
Serious Adverse Events (participants affected / at risk) | 0/91
Other Adverse Events (participants affected / at risk) | 8/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Large-group Transdiagnostic Course (N=86)
Temporary increase in anxiety or stress (Psychiatric disorders) | 3 (3) — self-reported, free text item
Other (Psychiatric disorders) | 6 (6) — self-reported, free text item

LIMITATIONS AND CAVEATS:
There was no control group, which implies that it is unclear if effects were causal. Patient satisfaction was not explored using qualitative methods.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT04522713/Prot_SAP_000.pdf